CLINICAL TRIAL: NCT00594204
Title: A 12-Week, Double-Blind, Randomized, Placebo-Controlled, Multicenter Study With Follow-Up Evaluating The Safety And Efficacy Of Varenicline Tartrate (CP-526,555-18) 1 Mg Bid For Smoking Cessation (Protocol A3051080)
Brief Title: Assessment of Safety and Efficacy of Varenicline in Patients That Wish to Stop Smoking
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3051080
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Results first posted 2010-07-05 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- varenicline (Active Comparator)
  Interventions: Drug: varenicline tartrate (CP-526, 555-18)
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: varenicline tartrate (CP-526, 555-18) — 1 mg twice a day for 12 weeks, starting with a 1-week titration period.
  Other Names: Chantix, Champix
  Arms: varenicline
Drug: Placebo — matching placebo 1 tablet twice a day for 12 weeks
  Arms: placebo

SUMMARY:
The primary objective of this protocol is to evaluate 12 weeks of treatment of varenicline compared to placebo for smoking cessation. Abstinence from cigarette smoking and other tobacco products (e.g., pipe, cigars, chew, snuff.) use during non-treatment follow-up period will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Current male or female cigarette smokers who are motivated to stop smoking.
* Smoked an average of 10 cigarettes per day during past year and the month prior to first visit.

Exclusion Criteria:

* Patients who have used a nicotine replacement product, bupropion, clonidine or notriptyline within the past 6 months.
* Patients currently with depression or diagnosed with depression in past 12 months.
* Past or present history of psychosis, panic disorder, or bipolar disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 593 (Actual)
Dates: Start 2008-04; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (40):
- Brazil (5):
  - Pfizer Investigational Site, Fortaleza, Ceará
  - Pfizer Investigational Site, Porto Alegre, Centro
  - Pfizer Investigational Site, Juiz de Fora, Minas Gerais
  - Pfizer Investigational Site, Botucatu, São Paulo
  - Pfizer Investigational Site, São Paulo, São Paulo
- Colombia (2):
  - Pfizer Investigational Site, Medellín, Antioquia
  - Pfizer Investigational Site, Barranquilla, Atlántico
- Pfizer Investigational Site, San Pedro, Provincia de San José, Costa Rica
- Pfizer Investigational Site, Cairo, Egypt, Egypt
- Pfizer Investigational Site, Amman, Jordan, Jordan
- Lebanon (2):
  - Pfizer Investigational Site, Beirut, Lebanon
  - Pfizer Investigational Site, Beirut Lebanon, Lebanon
- Mexico (3):
  - Pfizer Investigational Site, México, D.f.
  - Pfizer Investigational Site, Morelia, Michoacán
  - Pfizer Investigational Site, Monterrey, Nuevo León
- Saudi Arabia (2):
  - Pfizer Investigational Site, Jeddah
  - Pfizer Investigational Site, Riyadh
- South Africa (13):
  - Pfizer Investigational Site, Tygerberg, Cape Town
  - Pfizer Investigational Site, Bloemfontein, Free State
  - Pfizer Investigational Site, Benoni, Gauteng
  - Pfizer Investigational Site, Midrand, Gauteng
  - Pfizer Investigational Site, Pretoria, Gauteng
  - Pfizer Investigational Site, Soweto, Johannesburg
  - Pfizer Investigational Site, Durban, KwaZulu-Natal
  - Pfizer Investigational Site, Sydenham, Durban, KwaZulu-Natal
  - Pfizer Investigational Site, Hillcrest, Pretoria
  - Pfizer Investigational Site, Cape Town, Western Cape
  - Pfizer Investigational Site, Paarl, Cape Town, Western Cape
  - Pfizer Investigational Site, Durban
  - Pfizer Investigational Site, Lyttelton
- United Arab Emirates (6):
  - Pfizer Investigational Site, Dubai, United Arab Emirates
  - Pfizer Investigational Site, Abu Dhabi
  - Pfizer Investigational Site, Al Ain City
  - Pfizer Investigational Site, Dubai
  - Pfizer Investigational Site, Jumeirah/Dubai
  - Pfizer Investigational Site, Ras Al Khaima
- Venezuela (4):
  - Pfizer Investigational Site, Caracas, Distrito Federal
  - Pfizer Investigational Site, Barquisimeto, Lara
  - Pfizer Investigational Site, Gran Caracas, Miranda
  - Pfizer Investigational Site, Caracas

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Bolliger CT, Issa JS, Posadas-Valay R, Safwat T, Abreu P, Correia EA, Park PW, Chopra P. Effects of varenicline in adult smokers: a multinational, 24-week, randomized, double-blind, placebo-controlled study. Clin Ther. 2011 Apr;33(4):465-77. doi: 10.1016/j.clinthera.2011.04.013. PMID 21635992
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051080&StudyName=Assessment%20of%20safety%20and%20efficacy%20of%20varenicline%20in%20patients%20that%20wish%20to%20stop%20smoking%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Varenicline: 0.5 mg once daily (QD) for 3 days + 0.5 mg twice a day (BID) for 4 days, and then 1 mg BID for 11 weeks
- Placebo: matching placebo following the same treatment schema as the varenicline group
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 394 | 199
Received Treatment | 390 | 198
Completed | 336 | 154
Not Completed | 58 | 45
Not completed — Adverse Event | 15 | 3
Not completed — Lost to Follow-up | 9 | 5
Not completed — Withdrawal by Subject | 23 | 29
Not completed — Other | 4 | 3
Not completed — Lack of Efficacy | 3 | 4
Not completed — Randomized but not treated | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 390 | 198 | 588
Age, Customized [Number; unit: years]
  < 55 | 334 | 164 | 498
  55 - 65 | 49 | 28 | 77
  > 65 | 7 | 6 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165 | 68 | 233
  Male | 225 | 130 | 355

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Continuous Abstinence
Description: The number of participants who, at each contact from Week 9 through the given timepoint, reported no smoking and no use of other nicotine-containing products (Treatment Phase) or tobacco products (Nontreatment Phase) since the last study contact(on the Nicotine Use Inventory) and who did not have CO > 10 ppm
Time Frame: Weeks 9 through 24
Population: ITT
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 390 | 198
participants | 155 | 26
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — p-values are obtained from a logistic regression model including the main effects of treatment and country; Odds Ratio (OR) = 4.78, 95% CI [2.97 to 7.68] — Odds Ratios obtained from a logistic regression model including the main effects of treatment and country

2. Secondary Outcome: Number of Participants With Seven-day Point Prevalence of Abstinence
Description: Number of participants who, at the given visit or telephone contact, reported no smoking and no use of other nicotine-containing products (treatment phase) or tobacco products (non-treatment phase) in the last 7 days and who did not have CO >10 ppm on that day
Time Frame: Week 12 and 24
Population: ITT
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 390 | 198
participants
  Week 12 | 220 | 45
  Week 24 | 185 | 38
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Week 12; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — p-values obtained from a logistic regression model including the main effects of treatment and country; Odds Ratio (OR) = 5.0, 95% CI [3.3 to 7.5] — Odds ratios obtained from a logistic regression model including the main effects of treatment and country
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Week 24; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — p-values obtained from a logistic regression model including the main effects of treatment and country; Odds Ratio (OR) = 4.3, 95% CI [2.8 to 6.5] — Odds ratios obtained from a logistic regression model including the main effects of treatment and country

3. Primary Outcome: Number of Participants With 4-week Continuous Abstinence
Description: The number of participants who, at each visit from Week 9 through 12 (inclusive), reported no smoking and no use of other nicotine-containing products since the last study visit (on the Nicotine Use Inventory) and who did not have carbon monoxide (CO) > 10 parts per milion (ppm) at any of these visits
Time Frame: Weeks 9 through 12
Population: Intent-to-treat (ITT)
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 390 | 198
participants | 209 | 37
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; p-value are obtained from a logistic regression model including the main effects of treatment and country; Odds Ratio (OR) = 5.76, 95% CI [3.74 to 8.88] — Odds Ratios obtained from a logistic regression model including the main effects of treatment and country

ADVERSE EVENTS:
Arm/Group | Varenicline | Placebo
Serious Adverse Events (participants affected / at risk) | 11/390 | 2/198
Other Adverse Events (participants affected / at risk) | 224/390 | 82/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=390) | Placebo (N=198)
Bradycardia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Appendicectomy (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=390) | Placebo (N=198)
Abdominal pain (Gastrointestinal disorders) | 9 | 1
Abdominal pain upper (Gastrointestinal disorders) | 16 | 5
Constipation (Gastrointestinal disorders) | 23 | 10
Diarrhoea (Gastrointestinal disorders) | 9 | 2
Dry mouth (Gastrointestinal disorders) | 14 | 8
Dyspepsia (Gastrointestinal disorders) | 13 | 6
Flatulence (Gastrointestinal disorders) | 7 | 5
Nausea (Gastrointestinal disorders) | 103 | 16
Vomiting (Gastrointestinal disorders) | 12 | 1
Fatigue (General disorders) | 9 | 4
Irritability (General disorders) | 17 | 8
Malaise (General disorders) | 10 | 1
Bronchitis (Infections and infestations) | 9 | 4
Influenza (Infections and infestations) | 14 | 12
Nasopharyngitis (Infections and infestations) | 13 | 4
Upper respiratory tract infection (Infections and infestations) | 14 | 5
Increased appetite (Metabolism and nutrition disorders) | 9 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Dizziness (Nervous system disorders) | 13 | 9
Headache (Nervous system disorders) | 64 | 24
Somnolence (Nervous system disorders) | 16 | 9
Abnormal dreams (Psychiatric disorders) | 8 | 0
Anxiety (Psychiatric disorders) | 16 | 15
Depression (Psychiatric disorders) | 8 | 4
Drug dependence (Psychiatric disorders) | 3 | 5
Insomnia (Psychiatric disorders) | 50 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.